CLINICAL TRIAL: NCT02133781
Title: U19 Influenza Immunity: Protective Mechanisms Against a Pandemic Respiratory Virus. Project 1: B-cell Immunity to Influenza. Technical Development Project 1: Measuring the Immunome: Genomic Approaches to B-cell Repertoire- Year 1, 2009
Brief Title: B-cell Immunity to Influenza (SLVP017)- Year 1, 2009
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Cornelia L. Dekker, Professor, Pediatrics, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: SU-17218- 2009; 2U19AI057229-06 (NIH)
Record Dates: First submitted 2014-05-06; First posted 2014-05-08 (Estimated); Results first posted 2017-03-10 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-05

CONDITIONS: Influenza
Keywords: Inactivated influenza vaccine; Live, attenuated influenza vaccine; Child identical twins; Young and elderly adults
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Age 8-17 years (identical twins ) (Experimental): Participants will be randomized to receive either Fluzone® 2009-2010 Formula or FluMist® 2009-2010 Formula
  Interventions: Biological: Fluzone® 2009-2010 Formula; Biological: FluMist® 2009-2010 Formula
- Age 18-30 years (non-twins) (Experimental): Participants will be receive Fluzone® 2009-2010 Formula
  Interventions: Biological: Fluzone® 2009-2010 Formula
- Age >70 years (non-twins) (Experimental): Participants will receive Fluzone® 2009-2010 Formula
  Interventions: Biological: Fluzone® 2009-2010 Formula

INTERVENTIONS:
Biological: Fluzone® 2009-2010 Formula — This vaccine is given intramuscularly
  Other Names: Trivalent inactivated influenza vaccine (TIV); FDA-licensed seasonal influenza vaccine
Biological: FluMist® 2009-2010 Formula — This vaccine is given intranasally
  Other Names: Live, attenuated influenza vaccine (LAIV); FDA-licensed seasonal influenza vaccine
  Arms: Age 8-17 years (identical twins )

SUMMARY:
This is an exploratory study using a strategy that has not been previously employed to investigate the effects of age and vaccine type on specific kinds of immune responses to licensed, seasonal 2009-2010 influenza vaccines in children and adults.

DETAILED DESCRIPTION:
This study is being conducted in healthy male and female volunteers. 8-17 year-old identical twins will be randomly assigned to receive a single administration of the 2009-2010 formulation of either seasonal trivalent inactivated influenza vaccine (TIV) or live, attenuated influenza vaccine (LAIV). Twins within a pair will receive different vaccines. 18-30 year-old and 70-100 year-old subjects will receive a single administration of the 2009-2010 formulation of TIV. Blood samples to conduct the assays will be taken at pre-immunization, Day 7-8 and Day 28 post immunization.

ELIGIBILITY:
Inclusion Criteria:

* Otherwise healthy, ambulatory children 8-17 year-old twins, adults 18-30 years old (non-twin) or 70-100 year-old elderly non-twin adults.
* Willing to complete the informed consent process.
* Availability for follow-up for the planned duration of the study at least 28 days after immunization.
* Acceptable medical history by medical history and vital signs.

Exclusion Criteria:

* Prior off-study vaccination with the current seasonal TIV or LAIV in Fall 2009
* Allergy to egg or egg products, or to vaccine components, including gentamicin, gelatin, arginine or MSG (for LAIV only), or thimerosal (TIV multidose vials only).
* Life-threatening reactions to previous influenza vaccinations
* Asthma or history of wheezing (for volunteers randomized to LAIV)
* Active systemic or serious concurrent illness, including febrile illness on the day of vaccination
* History of immunodeficiency (including HIV infection)
* Known or suspected impairment of immunologic function, including, but not limited to, clinically significant liver disease, diabetes mellitus treated with insulin, moderate to severe renal disease, or any other chronic disorder which, in the opinion of the investigator, might jeopardize volunteer safety or compliance with the protocol.
* Blood pressure >150 systolic or >95 diastolic at first study visit
* Hospitalization in the past year for congestive heart failure or emphysema.
* Chronic Hepatitis B or C.
* Recent or current use of immunosuppressive medication, including systemic glucocorticoids (corticosteroid nasal sprays and topical steroids are permissible in all groups; inhaled steroid use is not permissible except for non-LAIV Group only). Use of oral steroids (<20 mg prednisone-equivalent/day) may be acceptable for volunteers 70-100 yrs of age after review by the investigator.
* Participants in close contact with anyone who has a severely weakened immune system should not receive LAIV
* Malignancy, other than squamous cell or basal cell skin cancer (includes solid tumors such as breast cancer or prostate cancer with recurrence in the past year, and any hematologic cancer such as leukemia).
* Autoimmune disease (including rheumatoid arthritis treated with immunosuppressive medication such as Plaquenil, methotrexate, prednisone, Enbrel) which, in the opinion of the investigator, might jeopardize volunteer safety or compliance with the protocol.
* History of blood dyscrasias, renal disease, or hemoglobinopathies requiring regular medical follow up or hospitalization during the preceding year
* Use of any anti-coagulation medication such as Coumadin or Lovenox, or anti-platelet agents such as aspirin (except up to 325 mg. per day), Plavix, or Aggrenox must be reviewed by investigator to determine if this would affect the volunteer's safety.
* Receipt of blood or blood products within the past 6 months
* Medical or psychiatric condition or occupational responsibilities that preclude participant compliance with the protocol
* Inactivated vaccine 14 days prior to vaccination
* Live, attenuated vaccine within 60 days of vaccination
* History of Guillain-Barré Syndrome
* Pregnant or lactating woman
* Use of investigational agents within 30 days prior to enrollment
* Donation of the equivalent of a unit of blood within 6 weeks prior to enrollment
* Any condition which, in the opinion of the investigator, might interfere with volunteer safety, study objectives or the ability of the participant to understand or comply with the study protocol.

Ages: 8 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2009-07; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cornelia L Dekker, MD, Principal Investigator — Stanford University; Harry B Greenberg, MD, Principal Investigator — Stanford University; Xiaosong He, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford LPCH Vaccine Program, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] He XS, Sasaki S, Narvaez CF, Zhang C, Liu H, Woo JC, Kemble GW, Dekker CL, Davis MM, Greenberg HB. Plasmablast-derived polyclonal antibody response after influenza vaccination. J Immunol Methods. 2011 Feb 28;365(1-2):67-75. doi: 10.1016/j.jim.2010.12.008. Epub 2010 Dec 21. PMID 21182843
- [Background] Sasaki S, Sullivan M, Narvaez CF, Holmes TH, Furman D, Zheng NY, Nishtala M, Wrammert J, Smith K, James JA, Dekker CL, Davis MM, Wilson PC, Greenberg HB, He XS. Limited efficacy of inactivated influenza vaccine in elderly individuals is associated with decreased production of vaccine-specific antibodies. J Clin Invest. 2011 Aug;121(8):3109-19. doi: 10.1172/JCI57834. Epub 2011 Jul 25. PMID 21785218
- [Background] He XS, Sasaki S, Baer J, Khurana S, Golding H, Treanor JJ, Topham DJ, Sangster MY, Jin H, Dekker CL, Subbarao K, Greenberg HB. Heterovariant cross-reactive B-cell responses induced by the 2009 pandemic influenza virus A subtype H1N1 vaccine. J Infect Dis. 2013 Jan 15;207(2):288-96. doi: 10.1093/infdis/jis664. Epub 2012 Oct 29. PMID 23107783
- [Background] Jiang N, He J, Weinstein JA, Penland L, Sasaki S, He XS, Dekker CL, Zheng NY, Huang M, Sullivan M, Wilson PC, Greenberg HB, Davis MM, Fisher DS, Quake SR. Lineage structure of the human antibody repertoire in response to influenza vaccination. Sci Transl Med. 2013 Feb 6;5(171):171ra19. doi: 10.1126/scitranslmed.3004794. PMID 23390249
- [Background] Brodin P, Jojic V, Gao T, Bhattacharya S, Angel CJ, Furman D, Shen-Orr S, Dekker CL, Swan GE, Butte AJ, Maecker HT, Davis MM. Variation in the human immune system is largely driven by non-heritable influences. Cell. 2015 Jan 15;160(1-2):37-47. doi: 10.1016/j.cell.2014.12.020. PMID 25594173
- [Derived] de Bourcy CFA, Dekker CL, Davis MM, Nicolls MR, Quake SR. Dynamics of the human antibody repertoire after B cell depletion in systemic sclerosis. Sci Immunol. 2017 Sep 29;2(15):eaan8289. doi: 10.1126/sciimmunol.aan8289. PMID 28963118

RESULTS

PARTICIPANT FLOW:
Groups:
- Age > 70 Years (Non-twins): Participants will receive Fluzone® 2009-2010 Formula
  Fluzone® 2009-2010 Formula: This vaccine is given intramuscularly
Period: Overall Study
Arm/Group | Age 8-17 Years (Identical Twins ) | Age 18-30 Years (Non-twins) | Age > 70 Years (Non-twins)
Started | 6 | 24 | 21
Completed | 6 | 24 | 21
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Age 8-17 Years (Identical Twins ) | Age 18-30 Years (Non-twins) | Age > 70 Years (Non-twins) | Total
Number analyzed (Participants) | 6 | 24 | 21 | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6 | 0 | 0 | 6
  Between 18 and 65 years | 0 | 24 | 0 | 24
  >=65 years | 0 | 0 | 21 | 21
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 16 | 11 | 33
  Male | 0 | 8 | 10 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 0 | 2
  Not Hispanic or Latino | 6 | 22 | 21 | 49
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 10 | 0 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 0 | 2
  White | 6 | 10 | 21 | 37
  More than one race | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 6 | 24 | 21 | 51

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants From Each Arm Who Received Influenza Vaccine
Time Frame: Day 0 to 28
Measure: Count of Participants; unit: Participants
Arm/Group | Age 8-17 Years (Identical Twins ) | Age 18-30 Years (Non-twins) | Age > 70 Years (Non-twins)
Number analyzed (Participants) | 6 | 24 | 21
Participants | 6 | 24 | 21

2. Secondary Outcome: Number of Participants With Related Adverse Events
Time Frame: Day 0 to 28 post-immunization
Measure: Count of Participants; unit: Participants
Arm/Group | Age 8-17 Years (Identical Twins ) | Age 18-30 Years (Non-twins) | Age > 70 Years (Non-twins)
Number analyzed (Participants) | 6 | 24 | 21
Participants | 0 | 0 | 0

3. Other Pre Specified Outcome: To Investigate the Effects of Age and Vaccine Type on B-cell Responses to Influenza Vaccine
Time Frame: Day 0 to 28
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Day 0 to Day 28 of study participation
Description: Clinical Assessment performed at each visit
Arm/Group | Age 8-17 Years (Identical Twins ) | Age 18-30 Years (Non-twins) | Age > 70 Years (Non-twins)
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/24 | 0/21
Other Adverse Events (participants affected / at risk) | 0/6 | 0/24 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No